CLINICAL TRIAL: NCT06568588
Title: Effects of Probiotic Consumption in Children With Autism Spectrum Disorder (ASD) in the Metropolitan District of Quito, Ecuador
Brief Title: Effects of Probiotic Consumption in Children With Autism Spectrum Disorder (ASD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad San Francisco de Quito (Other)
Collaborators: Biocodex (Industry); Neurodesarrollo Quito (Unknown); University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Paúl Cárdenas, PhD, Professor at the Institute of Microbiology, Universidad San Francisco de Quito
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023032
Record Dates: First submitted 2024-08-14; First posted 2024-08-23 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: intestinal microbiota; Intestinal metabolome; Autism spectrum disorder; ASD; Nutrition; Immune status; Gastrointestinal symptoms
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Children diagnosed with ASD will be randomly organized into 2 groups. Group A (n=33) will receive Sb supplements at a dose of 250 mg 3 times a day for a period of 4 months. While Group B (n=33) will not receive supplementation for 4 months. This will be followed by a 30-day "washout" period, during which time neither group consumes probiotics. After this time, the children's groups will change treatment for another four months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First four months with Sb (Group A) (Experimental): Children that receive Sb supplements in the initial 4 months of the study.
  Interventions: Drug: S. boulardii CNCM (National Collection of Cultures of Microorganisms) I-745
- Last four months with Sb (Group B) (Experimental): Children that receive Sb supplements in the final 4 months of the study.
  Interventions: Drug: S. boulardii CNCM (National Collection of Cultures of Microorganisms) I-745

INTERVENTIONS:
Drug: S. boulardii CNCM (National Collection of Cultures of Microorganisms) I-745 — 250 mg three times a day for 4 months
  Other Names: Floratil

SUMMARY:
The goal of this clinical trial is to determine the effects of Saccharomyces boulardii (Sb) consumption on Ecuadorian children with a diagnosis of autism spectrum disorder (ASD) and digestive symptoms. Saccharomyces boulardii is a probiotic, in other words, a beneficial microorganism. The main question it aims to answer is: Does Sb improve intestinal health, defenses against infections, nutrition and behavior of the participants. Researchers will compare children when they are taking and not taking Saccharomyces boulardii to know if there are changes in digestive symptoms, immune system function, nutritional status and behavior. Participants will take Saccharomyces boulardii for 4 months and will be 4 months without taking Sb. All participants must provide stool, urine and blood samples. A medical, nutritional and psychological team will follow the participants at least 5 times during the study.

DETAILED DESCRIPTION:
Autism Spectrum disorder (ASD), is a group of neurodevelopmental abnormalities that begin in early childhood, frequently characterized by problems in communication and social behavior. Metabolites produced by the gut microbiome may affect gastrointestinal (Gl) tract and central nervous system (CNS) functions supporting the presence of the gut- brain-axis. Previous studies have demonstrated changes in the intestinal microbiome in children with ASD compared with neurotypical controls. It is possible that dietary modifications, including the use of probiotics, in children with ASD could positively modify Gl and CNS functions. Few clinical studies have been carried out to assess the effects of probiotic consumption by children with ASD on their microbiota composition, intestinal function and behavior in developing countries. Consequently, the general objective of the study is to determine the effects of probiotics supplementation in gut microbiota composition, nutritional status and immune status in children with ASD.

A randomized crossover study will be conducted including children diagnosed with ASD, living within the Metropolitan District of Quito. After verifying the inclusion and exclusion criteria, 66 participants will be selected. Initially, children diagnosed with ASD will be randomly organized into 2 groups. Group A (n=33) will receive Sb supplements at a dose of 250 mg 3 times a day for a period of 4 months. While Group B (n=33) will not receive supplementation for 4 months. This will be followed by a 30-day "washout" period, during which time neither group consumes probiotics. After this time, the children's groups will change treatment for another four months. The investigators will analyze behavior, gut microbiome, metabolome, nutritional status and gastrointestinal symptoms to determine the changes caused by Sb consumption. Participants will be followed up at months 1, 4, 5, 9 10 of the study. At each follow-up, stool, blood and urine samples will be collected for the different analyzes.

A sociodemographic survey will be applied to determine the epidemiological parameters of the participants. The behavioral parameters of each child will be evaluated by means of psychological assessments. Tests that will be applied are: Autism Diagnostic Observation Schedule, Second Edition (ADOS- 2); Autism Diagnostic Interview-Revised (ADI-R); Wechsler Intelligence Scale for Children (WISC); Adaptive Behavior Assessment System (ABAS); Wechsler Preschool and Primary Scale of Intelligence (WPPSI); Battelle Developmental Inventory (BATELLE). For the evaluation of nutritional status, anthropometric measurements (weight, height, BMI) will be taken and percentiles and Z-scores will be calculated. In addition, a 24-hour recall questionnaire will be applied. Roma IV test will be applied to evaluate gastrointestinal symptoms. To determine the immunological status, the investigators will measure interleukins and growth factors in blood.

Regarding the analysis of the gut microbiota, the investigators will start with DNA extraction from stool samples. All raw sequences obtained from the Illumina sequencer will be analyzed to determine: taxonomic composition, alpha and beta diversity, functional annotation and differential microbial relative abundance between the two groups. Functional annotation will be performed using Human Microbiome Project Unified Metabolic Analysis Network (HumanN) software. Taxonomic assignment will be done using Metagenomic Phylogenetic Analysis (Metaphlan) software. Diversity metrics will be calculated using the Vegan diversity R package. To compare alpha diversity analysis, Chao 1, Shannon and Simpson's index will be calculated. For Beta diversity comparison, the Analysis of Ecological Data (ade4) function in the R package will be used to generate principal component analysis using Bray-Curtis, Jaccard, unweighted Unifrac and weighted Unifrac distance metrics. Linear discriminant analysis will be used in conjunction with the sample size effect measurement test (LEfSe) to perform differential microbial relative abundance analysis between the two groups.

The investigators will perform metabolome analysis on blood, fecal samples and urine. Metabolome assignment will be by 2D experiments based on signal in Proton nuclear magnetic resonance (H-NMR), using the human metabolome database and the biological magnetic resonance metabolome database.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Autistic Spectrum Disorders (ASD).
* History of gastrointestinal (GI) disorders, recurrent diarrhea, during the past 6 months.
* Children attending learning or therapy centers or schools.
* Age between 5 and 12 years of age.
* Children whose parents or guardians consent their participation in the study.
* Children who can provide the required biological samples, and their guardians must provide the necessary information to complete the established instruments.
* The parents or guardians of the children must sign the informed consent form in order to be part of the study.

Exclusion Criteria:

* Use of antibiotics, systemic steroids or antifungal medication during the last 15 days prior to fecal sample collection.
* Acute gastrointestinal, respiratory or febrile processes.
* Severe chronic comorbidities such as cancer, immunosuppression, obstructive respiratory disorders, Crohn's disease, ulcerative colitis, among others, at the discretion of the investigators.
* Probiotics consumption in the last three months prior to study enrollment.
* History of allergy or hypersensitivity to Saccharomyces boulardii or its components, or allergy to yeasts.
* Contraindication and special warning to Saccharomyces boulardii according to the technical Data Sheets, including central venous catheter carriers.
* Simultaneous participation in clinical studies, or in exclusion periods of a previous clinical study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2024-01-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Modifications of gastrointestinal symptoms during Sb administration | Gastrointestinal symptoms will be evaluated monthly, through study completion, an average of 1 year
  Changes in gastrointestinal symptoms of children with ASD when they are receiving Sb. Symptoms will be evaluated with Rome IV Pediatric Questionnaire Parent Report For Children and Adolescents Age 4+.
Modifications of gastrointestinal microbiota during Sb administration | Fecal samples will be analyzed at months 1, 4, 5, 9 and 10 of the study.
  Changes in alpha diversity, beta diversity, taxonomic composition, functional annotation and differential microbial relative abundance of gastrointestinal microbiota of children with ASD when they are receiving Sb supplementation.
Modifications of fecal metabolome during Sb administration | Fecal samples will be analyzed at months 1, 4, 5, 9 and 10 of the study.
  Changes in the fecal metabolome of children with ASD when they are receiving Sb supplementation. Metabolome will be determined with 2D experiments based on signals in H-NMR, using the human metabolome database and the biological magnetic resonance metabolome database.
Modifications of blood metabolome during Sb administration | Blood samples will be analyzed at months 1, 4, 5, 9 and 10 of the study.
  Changes in blood metabolome of children with ASD when they are receiving Sb supplementation. Metabolome will be determined with 2D experiments based on signals in H-NMR, using the human metabolome database and the biological magnetic resonance metabolome database.
Modifications of urine metabolome during Sb administration | Urine samples will be analyzed at months 1, 4, 5, 9 and 10 of the study.
  Changes in urine metabolome of children with ASD when they are receiving Sb supplementation. Metabolome will be determined with 2D experiments based on signals in H-NMR, using the human metabolome database and the biological magnetic resonance metabolome database.
Modifications of body mass index (BMI) during Sb administration | BMI will be determined at months 1, 4, 5, 9 and 10 of the study.
  Changes in the BMI of children with ASD when they are receiving Sb supplementation. To obtain BMI, weight (in kilograms) and height (in meters) will be measured.
Modifications of nutrient intake during Sb administration | Nutrient intake will be determined at months 1, 4, 5, 9 and 10 of the study.
  Changes in the nutrient intake of children with ASD when they are receiving Sb supplementation. The 24-hour reminder questionnaire will be applied to quantify nutrient intake.
Modifications of immune function during Sb administration | Blood samples for interleukins and growth factors determination will be analyzed at months 1,4, 5, 9,10 of the study
  Changes in the immune function of children with ASD when they are receiving Sb supplementation. Levels of interleukins and growth factors will be determined. Specifically, interleukin(IL)-1, IL-4, IL-6, IL-8, tumoral necrosis factor (TNF) -α, interferon (IFN)-γ, IL-10, transforming growth factor (TGF)-β will be measured.
Modifications of behavior during Sb administration | ADOS-2 test will be performed at months 1, 4, 5, 9, 10 of the study.
  Changes in the behavior of children with ASD when they are receiving Sb supplementation. ADOS- 2 test will be applied to determine conduct in different situations, sensory response and adaptive functioning. The total scores range from 15 to 60, and a higher score means a worse outcome.
Modifications in the intelligence levels during Sb administration | Tests will be performed at months 1, 4, 5, 9, 10 of the study.
  Changes in the intelligence levels of children with ASD when they are receiving Sb supplementation. Different tests will be used according to the age and language level of the participants. WISC will be used on children from 7 years 4 months of age. WPPSI will be applied to children 7 years 3 months or younger. BATTELLE will be used for children 8 years old or younger who have a low language level. With all of these tests, a higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Paúl A Cárdenas, PhD, Principal Investigator — Universidad San Francisco de Quito
Locations (1):
- Neurodesarrollo Quito, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification.
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] De Angelis M, Francavilla R, Piccolo M, De Giacomo A, Gobbetti M. Autism spectrum disorders and intestinal microbiota. Gut Microbes. 2015;6(3):207-13. doi: 10.1080/19490976.2015.1035855. PMID 25835343
- [Background] Slattery J, MacFabe DF, Frye RE. The Significance of the Enteric Microbiome on the Development of Childhood Disease: A Review of Prebiotic and Probiotic Therapies in Disorders of Childhood. Clin Med Insights Pediatr. 2016 Oct 9;10:91-107. doi: 10.4137/CMPed.S38338. eCollection 2016. PMID 27774001
- [Background] Zurita MF, Cardenas PA, Sandoval ME, Pena MC, Fornasini M, Flores N, Monaco MH, Berding K, Donovan SM, Kuntz T, Gilbert JA, Baldeon ME. Analysis of gut microbiome, nutrition and immune status in autism spectrum disorder: a case-control study in Ecuador. Gut Microbes. 2020 May 3;11(3):453-464. doi: 10.1080/19490976.2019.1662260. Epub 2019 Sep 18. PMID 31530087
- [Background] Srikantha P, Mohajeri MH. The Possible Role of the Microbiota-Gut-Brain-Axis in Autism Spectrum Disorder. Int J Mol Sci. 2019 Apr 29;20(9):2115. doi: 10.3390/ijms20092115. PMID 31035684